CLINICAL TRIAL: NCT01305941
Title: A Phase II Study Evaluating The Efficacy And Tolerability Of Everolimus (RAD001) In Combination With Trastuzumab And Vinorelbine In The Treatment Of Progressive HER2-Positive Breast Cancer Brain Metastases
Brief Title: A Study Of Everolimus, Trastuzumab And Vinorelbine In HER2-Positive Breast Cancer Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1025; 11-0242 (Other: UNC IRB assigned protocol number)
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: HER-2 Positive Breast Cancer
Keywords: everolimus; trastuzumab; vinorelbine; RAD001; Breast Cancer; Herceptin; Navelbine; Lineberger Comprehensive Cancer Center; Brain Metastases
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — Everolimus; Vinorelbine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus +Vinorelbine + trastuzumab (Experimental): daily everolimus plus weekly (Days 1, 8, and 15) vinorelbine and trastuzumab
  Interventions: Drug: Everolimus; Drug: Vinorelbine; Drug: Trastuzumab

INTERVENTIONS:
Drug: Everolimus — everolimus 5 mg PO daily as two 2.5-mg tablets
  Other Names: RAD001
Drug: Vinorelbine — vinorelbine 25 mg/m2 will be administered via IV infusion over 6-10 minutes weekly.
  Other Names: Navelbine
Drug: Trastuzumab — 2 mg/kg IV administered over 30 minutes weekly
  Other Names: Herceptin

SUMMARY:
Purpose: This study is a single-arm, open-label phase II clinical trial testing the hypothesis that daily everolimus plus weekly vinorelbine and trastuzumab will be effective, safe, and tolerable among patients with human epidermal growth factor receptor 2 (HER2)-positive breast cancer brain metastases. Once enrolled, patients will receive everolimus PO daily in combination with weekly intravenous (IV) vinorelbine and trastuzumab. Cycles will be repeated every 3 weeks (21 days). At the time of progression, patients will come off study.

Participants: Up to 35 adults over 21 with HER-2 positive breast cancer that has metastasized to the brain.

DETAILED DESCRIPTION:
STUDY OBJECTIVES Primary Objective -To determine the intracranial objective response rate of mTOR inhibition (everolimus) in combination with vinorelbine and trastuzumab in the treatment of HER2-positive, progressive breast cancer brain metastases as defined via modified RECIST criteria.

Secondary Objectives

* To determine the intracranial objective response rate of mechanistic target of rapamycin (mTOR) inhibition (everolimus) in combination with vinorelbine and trastuzumab in the treatment of HER2-positive, progressive breast cancer brain metastases as defined by MacDonald criteria.
* To evaluate the safety and tolerability of everolimus in combination with trastuzumab and vinorelbine as assessed via the NCI CTCAE version 4.0
* To evaluate time to intracranial progression after administration of everolimus in combination with trastuzumab and vinorelbine as defined via modified RECIST criteria
* To evaluate the extracranial objective response rate as determined by RECIST 1.1 criteria after administration of everolimus in combination with trastuzumab and vinorelbine.
* To evaluate the extracranial time to progression as determined by RECIST 1.1 criteria after administration of everolimus in combination with trastuzumab and vinorelbine.
* To evaluate progression free survival (PFS) and overall survival (OS) after administration of everolimus in combination with trastuzumab and vinorelbine.
* To evaluate the impact of everolimus in combination with trastuzumab and vinorelbine on quality of life as measured by the Functional Assessment of Cancer Therapy Breast (FACT-B) and Functional Assessment of Cancer Therapy Brain (FACT-Br) questionnaires.

Exploratory Objective

-To evaluate biomarkers in archival tumor tissue samples and correlate with therapeutic response to everolimus in combination with vinorelbine and trastuzumab.

Following Hepatitis B antiviral prophylaxis if required, or following screening and informed consent if antiviral therapy is not needed, treatment will be initiated with everolimus PO daily in combination with weekly intravenous (IV) vinorelbine and trastuzumab (Days 1, 8, and 15)

A cycle is defined as 3 weeks (21 days). Cycles of therapy will be repeated until documented disease progression, unacceptable toxicity, or patient withdrawal from study for other reasons, including death.

ELIGIBILITY:
Inclusion Criteria

* Histologically-confirmed HER2-positive (IHC 3+ or fluorescence in situ hybridization (FISH) amplified; by clinical assay on either primary or metastatic tumor) adenocarcinoma of the breast with at least one progressive and/or new metastatic brain lesion (>/=5 mm on radiographic imaging) after receipt of intracranial radiation therapy (whole brain radiation therapy, stereotactic radiosurgery, gamma knife, or equivalent). Patients in whom brain metastases (BM) are asymptomatic and detected during routine brain MRI screening per institutional protocols are eligible.
* Prior intracranial radiation therapy (whole brain radiation therapy, stereotactic radiosurgery, gamma knife or equivalent) is allowed but not required.
* Patients with no prior treatment with intracranial Response (ICR) may be included unless ICR is emergently indicated (in consultation with a local therapist, ie neurosurgeon or radiation oncologist)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy >12 weeks.
* At least 21 years of age.
* No prior mTOR inhibitors
* Prior navelbine allowed provided navelbine therapy discontinued >/= 12 months from Day 1 of treatment under this protocol.
* Last anti-cancer treatment (including any investigational drug) >/= 2 weeks from initiation of protocol based therapy, provided all adverse events (AEs) (other than alopecia) have resolved to ≤grade 1 at baseline.
* No active serious infection or other comorbid illness which would impair ability to participate in the trial.
* Left ventricular ejection fraction assessment (echocardiogram or multigated acquisition scan (MUGA) scan) performed within 4 weeks prior to study initiation, showing a Left ventricular ejection fraction (LVEF) value ≥ lower limit of normal (LLN).
* If patient is on dexamethasone, must be on stable or decreasing dose of dexamethasone for ≥7 days. If patient is on different glucocorticoid e.g., prednisone, must be converted to dexamethasone prior to enrollment. Refer to dose modification of everolimus for patients taking dexamethasone.
* Interval ≥4 weeks between open brain biopsy and initiation of protocol-based therapy.
* international normalized ratio (INR) ≤2.0. Anticoagulation is allowed if target INR ≤2.0 on a stable dose of warfarin or if patient on a stable dose of Low-molecular-weight (LMW) heparin for >1 weeks at time of enrollment.
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤2.5 x ULN. Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Patients must have adequate organ function as evidenced by:
* Absolute neutrophil count ≥1.5/µL
* Platelet count ≥100,000/µL
* Hg ≥9 g/dL
* Bilirubin ≤1.5 x upper limit of normal (ULN)
* aspartate aminotransferase (AST) or Alanine transaminase (ALT) ≤2.5 x ULN (≤5 x ULN if liver metastases are present)
* Serum creatinine ≤1.5 x ULN
* Archived, paraffin-embedded tissue block (primary or metastatic) available for genomic studies is required.
* Signed, institutional review board (IRB)-approved written informed consent.

Exclusion Criteria

* Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus); patients who have received prior treatment with navelbine within prior 12 months.
* patients with a known hypersensitivity to everolimus or other rapamycins (e.g. sirolimus, temsirolimus) or to its excipients.
* Patients requiring treatment with any other systemic glucocorticoid. Note: This restriction regarding choice of glucocorticoid does not apply should patient need <2 week course of glucocorticoid for treatment of non-infectious pneumonitis during study (see section 4.5.2).
* Patients with a known hypersensitivity to vinorelbine or to its excipients.
* Prior allergic reaction to trastuzumab for the treatment of metastatic breast cancer.
* Concurrent or planned radiation, hormonal, chemotherapeutic, experimental or targeted biologic therapy.
* Peripheral neuropathy ≥grade 3.
* Evidence of frank hemorrhage or impending herniation on baseline brain imaging. Note: asymptomatic micro-hemorrhage is allowed.
* Evidence of diffuse leptomeningeal disease on brain MRI or by previously documented Cerebrospinal fluid (CSF) cytology. Note: discrete dural metastases are permitted.
* Active cardiac disease including any of the following:

  * Angina pectoris that requires the use of anti-anginal medication;
  * Ventricular arrhythmias except for benign premature ventricular contractions;
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication;
  * Conduction abnormality requiring a pacemaker;
  * Valvular disease with documented compromise in cardiac function;
  * Symptomatic pericarditis
* History of cardiac dysfunction including any one of the following:

  * Myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function;
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV);
  * Documented cardiomyopathy
* Patients who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia), or patients that may require major surgery during the course of the study.
* Patients should not receive immunization with attenuated live vaccines within 1 week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella, and Typhoid Vaccine Live Oral (TY21a) typhoid vaccines.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * severely impaired lung function, defined as spirometry and diffusion lung capacity for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is ≤88% at rest on room air
  * uncontrolled diabetes, defined as fasting serum glucose >1.5 x ULN (Note: Optimal glycemic control should be achieved before starting trial therapy)
  * active (acute or chronic) or uncontrolled severe infections
  * liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).

Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B Virus (HBV) DNA and hepatitis C Virus (HCV) RNA polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.

* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low-dose warfarin and aspirin or equivalent, as long as the INR ≤2.0).
* Unable or unwilling to discontinue use of prohibited fruit (or its juices) and prohibited medications listed in Appendices II and III for at least 14 days or 5 half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Female patients who are pregnant or breastfeeding, or adults of reproductive potential who are not using effective birth control methods. Adequate contraception must be used throughout the trial and for 8 weeks after the last dose of study drug, by both sexes. Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test within 7 days prior to everolimus initiation.
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
* Contraindication to gadolinium-enhanced MRI imaging.
* Inability to comply with study and/or follow-up procedures.
* History of noncompliance to medical regimens.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2016-08 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey K Anders, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University Of Alabama at Birmingham, Birmingham, Alabama
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Van Swearingen AED, Siegel MB, Deal AM, Sambade MJ, Hoyle A, Hayes DN, Jo H, Little P, Dees EC, Muss H, Jolly T, Zagar TM, Patel N, Miller CR, Parker JS, Smith JK, Fisher J, Shah N, Nabell L, Nanda R, Dillon P, Abramson V, Carey LA, Anders CK. LCCC 1025: a phase II study of everolimus, trastuzumab, and vinorelbine to treat progressive HER2-positive breast cancer brain metastases. Breast Cancer Res Treat. 2018 Oct;171(3):637-648. doi: 10.1007/s10549-018-4852-5. Epub 2018 Jun 25. PMID 29938395
- See also: Lineberger Comprehensive Cancer Center — http://cancer.med.unc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 institutions between September, 2011 and May, 2016.
Pre-assignment Details: A total of 41 patients were consented to this study. Of these, 6 patients were found ineligible, 2 withdrew prior to treatment, and 1 patient has disease progression prior to protocol therapy. Therefore only 32 patients were enrolled and participated in the trial.
Period: Overall Study
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Started | 32
Completed | 22
Not Completed | 10
Not completed — Adverse Event | 6
Not completed — Clinical decline | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 53 [28 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
Stage at breast cancer diagnosis [Count of Participants; unit: Participants] — Anatomic stage for NSCLC is the American Joint Committee on Cancer (AJCC) tumor, node, and metastases (TNM) system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced.
  Participants
    0-III | 19
    IV | 13
Median time since first brain metastases (years) [Median (Full Range); unit: years] | 1.12 [0.4 to 6.5]
Prior Systemic Chemotherapy (metastatic) [Count of Participants; unit: Participants] — Number of participants who received prior systemic chemotherapy.
  Participants | 30
Prior metastatic chemotherapy lines, # (range) [Median (Full Range); unit: Metastatic Lines] | 2 [0 to 7]
Prior anti-Her2 (metastatic) Agents [Count of Participants; unit: Participants]
  Trastuzumab | 29
  Lapatinib | 22
  Pertuzumab | 12
  Trastuzumab Emtansine (TDM-1) | 8
Prior Central Nervous System Local Therapy [Count of Participants; unit: Participants]
  Surgery | 10
  Whole brain radiation therapy | 22
  Stereotactic Radiosurgery (SRS) | 17
Recursive Partitioning Analysis (RPA) Score [Count of Participants; unit: Participants] — Recursive partitioning creates a decision tree that classifies members of a population by splitting it into sub-populations based on several dichotomous independent variables. The process is termed recursive because each sub-population may in turn be split an indefinite number of times.
  This includes three classes: Class 1 (patients <65 years, ECOG Performance Status of 0-1, controlled primary tumor, and no extracranial metastases), Class 3 (ECOG Performance Status of 2 or greater), and Class 2 (all others);
  Participants
    Class 1 | 10
    Class 2 | 21
    Class 3 | 1
Steroid use at baseline [Count of Participants; unit: Participants] — Treatment with corticosteroid drugs to reduce swelling, pain, and other symptoms of inflammation.
  Participants | 10
Extracranial disease at enrollment [Count of Participants; unit: Participants] — Outside of the cranium (bones that surround the brain).
  Participants | 20

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Objective Response Rate- Modified RECIST Criteria
Description: response will be evaluated via gadolinium-enhanced brain MRI using modified RECIST criteria.
  Complete Response (CR) - Disappearance of all target and nontarget lesions
  Partial Response (PR) - at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum longest diameter AND an absolute decrease of at least 5mm in at least one target lesion.
  Stable Disease (SD) - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameter since the treatment started.
  Progressive Disease (PD) - at least a 20% increase in the sum LD of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started AND an absolute increase in size of at least 5 mm in at least one target lesion OR the appearance of one or more new lesions of at least 6 mm in size.
Time Frame: 3 years
Population: Six subjects were not evaluable for response because there was no follow-up disease assessment done due to poor clinical status of subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 26
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 17
  Progressive Disease | 8

2. Secondary Outcome: Intracranial Response Rate- MacDonald Criteria
Description: Intracranial tumor lesions were evaluated via gadolinium-enhanced brain MRI using the MacDonald criteria. Measurable disease is defined as at least 1 measurable brain lesion accurately measured in at least 2 dimensions (longest diameter) as ≥5.0 mm. Tumor size is the product of the 2 longest bi-dimensional lines.
  Complete Response (CR)- Disappearance of all tumor on consecutive CT or MRI scans at least 1 month apart, off steroids for treatment of neurological symptoms, and neurologically stable or improved.
  Partial Response (PR)- ≥50% reduction in size of tumor on consecutive CT or MRI scans at least 1 month part, steroids stable or reduced, and neurologically stable or improved.
  Progressive Disease (PD)- ≥25% increase in size of tumor or any new tumor on CT or MRI scans, or neurologically worse, and steroids stable or increased due to neurologic symptoms.
  Stable Disease (SD)- all other situations Overall Response Rate (ORR) is the sum of partial responses (PRs) and CRs.
Time Frame: 3 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 26
Participants | 1

3. Secondary Outcome: Toxicity
Description: Grade 3 or higher toxicities of interest are reported. Toxicity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
  The NCI CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 32
Participants
  Alkaline phosphatase increased | 1
  Anemia | 5
  Anorexia | 1
  Asparate Aminotransferase Increased | 2
  Diarrhea | 1
  Febrile Neutropenia | 2
  Hyperkalemia | 1
  Lymphocyte Count Decreased | 3
  Mucositis Oral | 5
  Neutrophil Count Decreased | 13
  Pneumonitis | 1
  Sepsis | 3
  White Blood Cell Decreased | 11

4. Secondary Outcome: Time to Intracranial Progression.
Description: Time to intracranial progression after administration of everolimus in combination with trastuzumab and vinorelbine as defined via modified RECIST criteria.
  Progressive Disease (PD) - at least a 20% increase in the sum LD of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started AND an absolute increase in size of at least 5 mm in at least one target lesion OR the appearance of one or more new lesions of at least 6 mm in size.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 32
months | 3.93 [2.27 to 5.00]

5. Secondary Outcome: Extracranial Response
Description: Extracranial response was measured using RECIST 1.1 criteria and defined as the number of subjects achieving CR or PR.
  Complete Response (CR) - Disappearance of all target and nontarget lesions Partial Response (PR) - at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum longest diameter AND an absolute decrease of at least 5mm in at least one target lesion.
  Stable Disease (SD) - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameter since the treatment started.
  Progressive Disease (PD) - at least a 20% increase in the sum LD of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started AND an absolute increase in size of at least 5 mm in at least one target lesion OR the appearance of one or more new lesions of at least 6 mm in size.
Time Frame: 3 years
Population: Seven subjects were not evaluable for extra-cranial response because there was no follow-up disease assessment done due to poor clinical status of subjects. An additional 12 subjects were excluded since they did not have extra-cranial disease at baseline and one additional subject was non compliant for follow-up scans.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 12
Participants | 5

6. Secondary Outcome: Extracranial Time to Progression
Description: To evaluate the extracranial time to progression as determined by RECIST 1.1 criteria after administration of everolimus in combination with trastuzumab and vinorelbine.
  Progressive Disease (PD) - at least a 20% increase in the sum LD of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started AND an absolute increase in size of at least 5 mm in at least one target lesion OR the appearance of one or more new lesions of at least 6 mm in size.
Time Frame: 3 years
Population: Seven subjects were not evaluable for extra-cranial response due to no follow-up disease assessments due to poor clinical status; 12 subjects were excluded since they did not have extra-cranial disease at baseline; 1 subject was non compliant for follow-up scans; and 1 subject was excluded due to intracranial progression prior to extracranial.
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 6
months | 4.01 [1.97 to 8.26]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) after administration of everolimus in combination with trastuzumab and vinorelbine
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 32
years | 1.01 [.57 to 1.78]

8. Secondary Outcome: Functional Assessment of Cancer Therapy- Brain (FACT-Br) Change From Baseline to Assess Impact of Everolimus in Combination With Trastuzumab and Vinorelbine on Quality of Life
Description: The FACT-Br is a 23-question self-report questionnaire subscale administered with the Functional Assessment of Cancer Therapy- General (FACT-G) which contains concerns relevant to patients with brain tumors . Each question has a value 0-4. For some questions a higher indicates better outcome and others are the opposite. The former are summed as is, the latter are reversed in value before adding, such that each domain ranges from 0 to 4 times the number of questions in the domain, with 0 indicating worst and the highest possible value indicating best outcome. Total scores on the FACT-Br subscale range from 0 to 92 with lower scores indicating declining quality of life. The change from baseline is the difference in scores between the baseline and 9 week assessments.
Time Frame: 9 weeks
Population: Quality of life was an optional assessment for patients, so results are only reported for subjects who completed questionnaires at each timepoint
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 9
units on a scale | -1.0 [-5.0 to 4.8]

9. Secondary Outcome: Functional Assessment Cancer Therapy- Breast (FACT-B) From Baseline to 9 Weeks of Treatment to Assess Impact of Everolimus in Combination With Trastuzumab and Vinorelbine on Quality of Life
Description: The FACT-B is a 10-question self-report questionnaire subscale administered with the Functional Assessment of Cancer Therapy- General (FACT-G) which contains concerns relevant to patients with breast cancer. Each question has a value 0-4. For some questions a higher indicates better outcome and others are the opposite. The former are summed as is, the latter are reversed in value before adding, such that each domain ranges from 0 to 4 times the number of questions in the domain, with 0 indicating worst and the highest possible value indicating best outcome. Total scores on the FACT-B subscale range from 0 to 40 with lower scores indicating declining quality of life. The change from baseline is the difference in scores between the baseline and 9 week assessments.
Time Frame: 9 weeks
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
Number analyzed (Participants) | 11
units on a scale | 1.0 [-2.0 to 3.0]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Everolimus +Vinorelbine + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 29/32
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus +Vinorelbine + Trastuzumab (N=32)
Adrenal Insufficiency (Endocrine disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Creatinine Increased (Investigations) | 2
Fever (General disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion related reaction (General disorders) | 1
Laryngeal Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infection (Infections and infestations) | 1
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 2
Sepsis (Infections and infestations) | 3
Tremor (Nervous system disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus +Vinorelbine + Trastuzumab (N=32)
Abdominal pain (Gastrointestinal disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 10
Anxiety (Psychiatric disorders) | 3
Aspartate aminotransferase increased (Investigations) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3
Blood bilirubin increased (Investigations) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 3
Depression (Psychiatric disorders) | 5
Diarrhea (Gastrointestinal disorders) | 8
Dizziness (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Eye Disorders - Other, Specify (Eye disorders) | 2 — Verbatim: Dry eyelids; Eye muscle twitching
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Flu like symptoms (General disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypertension (Vascular disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 5
Infections And Infestations - Other, Specify (Infections and infestations) | 2 — Verbatim:infection to right thumb - laceration; folliculitis - facial; Right groin - sebaceous cyst or tiny abcess
Insomnia (Psychiatric disorders) | 6
Lymphocyte count decreased (Investigations) | 6
Memory impairment (Nervous system disorders) | 2
Mucosal infection (Infections and infestations) | 2
Mucositis oral (Gastrointestinal disorders) | 21
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal And Connective Tissue Disorder - Other, Specify (Musculoskeletal and connective tissue disorders) | 6 — Verbatim:Muscle cramps; muscle spasms-hands; Back muscle spasms; Cramping of feet and hands;Hand and jaw cramping; cramping legs
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Neutrophil count decreased (Investigations) | 17
Pain (General disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Papulopustular rash (Infections and infestations) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 9
Platelet count decreased (Investigations) | 7
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Respiratory, Thoracic And Mediastinal Disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 2 — Verbatim: Rhinorrhea; Nasal drainage clear, sometimes small amounts of blood
Skin And Subcutaneous Tissue Disorders - Other, Specify (Skin and subcutaneous tissue disorders) | 2 — Verbatim: Contact Dermatitis Bilateral Hands; Dermatitis (earlobes); blepharitis left eyelid
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 8
Vomiting (Gastrointestinal disorders) | 4
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days